CLINICAL TRIAL: NCT05930223
Title: Intravenous VAL-1221 Lafora Expanded Access Protocol (LEAP)
Brief Title: Intravenous VAL-1221 Lafora Expanded Access Protocol
Acronym: LEAP
Status: Available | Type: Expanded Access
Sponsor: Parasail, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: VAL1221-LEAP-01
Record Dates: First submitted 2023-06-25; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Lafora Disease
Keywords: Glycogen Storage Diseases; Polyglucosan Disorders; Progressive Myoclonic Epilepsy
MeSH Terms: conditions — Lafora Disease; Glycogen Storage Disease; Myoclonic Epilepsies, Progressive

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: VAL-1221 — VAL-1221 20mg/kg intravenous (IV) infusion every other week

SUMMARY:
Only qualified physicians treating a Lafora Disease patient may request VAL-1221 Expanded Access treatment under the Parasail Lafora Expanded Access Protocol (LEAP). According to FDA guidance, this protocol can enroll up to 10 patients. However, individual patient inclusion will ultimately be dependent on protocol eligibility, site geography, treatment requirements, and available supply of the investigational therapy. Inquiring physicians can submit a request by contacting the Central Contact personnel listed below in Contacts/Locations.

ELIGIBILITY:
Inclusion Criteria:

* Documented genetic diagnosis of Lafora Disease (LD) based on likely pathogenic or pathogenic variants in both alleles of either the EPM2A or the EPM2B gene
* Mid-stage in evolution of LD between 12 and 28 years of age
* Able and willing to comply with the protocol, including travel to Protocol Center, procedures, measurements and visits, including:

  * Adequately supportive psychosocial circumstances, in the opinion of the Investigator
  * Caregiver/trial partner committed to facilitate patient's involvement in the study who is reliable, competent, at least 18 years of age

Exclusion Criteria:

* Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the participant unsafe for inclusion or could interfere with the participant participating in or completing the protocol

Ages: 12 Years to 28 Years | Sex: All
Age Groups: Child, Adult